CLINICAL TRIAL: NCT00540904
Title: Prevention of Contrast Induced Nephropathy in Oncology Patients With Sodium Bicarbonate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-Silva
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2014-03-03 (Estimated); Status verified 2014-02

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: contrast; nephropathy; bicarbonate; prevention
MeSH Terms: conditions — Kidney Diseases | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sodium bicarbonate (Active Comparator): Solution 154 mEq/L of sodium bicarbonate
  Interventions: Drug: sodium bicarbonate
- Sodium chloride (Active Comparator): Solution of 154 mEq/L of NaCl
  Interventions: Drug: NaCl

INTERVENTIONS:
Drug: sodium bicarbonate — IV 154 mEq/L sodium bicarbonate. Infusion of 3 cc/Kg/h 1 hour before the injection of contrast and 1 cc/Kg/h after the injection.
  Arms: sodium bicarbonate
Drug: NaCl — IV 154 mEq/L solution of NaCl 0.9%. Infusion of 3 cc/Kg/h 1 hour before the injection of contrast and 1 cc/Kg/h after the injection.
  Arms: Sodium chloride

SUMMARY:
Contrast induced nephropathy is a rising cause of acute renal failure in all patients. A study published in JAMA 2004, show a superiority of a hydratation with sodium bicarbonate in comparison with the same volume hydratation with sodium bicarbonate. The investigators will try following the original protocol making 2 randomized groups of patients, with cancer diagnosis, >18 years old, with a GFR <60 and >30 ml/min/1,73m2 by MDRD formula and/or diabetic patients. In the group 1 the patients will receive a solution with 154 mEq/L of a sodium bicarbonate, 3 cc/Kg/h at 1 hour before the injection of contrast and 1 cc/Kg/h during and 6 hours before the injection. The primary end point will be the rise of 25% or more in creatinine or dialysis needed.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* cancer diagnosis
* GFR < 60 and > 30 ml/min/1,73m2 by MDRD formula or diabetic
* CT with contrast

Exclusion Criteria:

* dialysis needed
* uncontrolled hypertension
* changes in serum creatinine levels of at least 0.5 mg/dl during the previous 24 hours of procedure
* recent exposure to radiographic contrast agents (within previous two days of the study)
* administration of dopamine, mannitol , fenoldopam or N-Acetyl Cystein during the intended time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Development of contrast-induced nephropathy, defined as an increase in serum creatinine of 25% or more within 2 day after administration of contrast or dialysis needed | 2 days

SECONDARY OUTCOMES:
change in serum bicarbonate change in serum potassium change in serum glucose change in serum creatinine change in estimated glomerular filtration rate incidence of contrast induced nephropathy comparison of cholesterol level | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo G Silva, MD, Principal Investigator — Hospital do Cancer de Barretos - Fundação PIO XII
Locations (1):
- Hospital do Cancer de Barretos - Fundação PIO XII, Barretos, São Paulo, Brazil

REFERENCES:
- [Result] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204